CLINICAL TRIAL: NCT04753346
Title: Comparison of Cardiopulmonary Fitness Level With Normal Values After COVID-19 and Investigation of Factors Affecting Physical Capacity
Brief Title: Comparison of Cardiopulmonary Fitness Level With Normal Values After COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Burak Kamil Turan, MD, Ankara University
Other Study IDs: I11-670-20
Record Dates: First submitted 2021-02-12; First posted 2021-02-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: COVID 19
Keywords: Cardiopulmonary exercise test; Exercise capacity; COVID 19; 6 minute walk test
MeSH Terms: conditions — COVID-19 | interventions — Respiratory Function Tests; Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Mild Disease: Symptomatic patients meeting the case definition for COVID-19 without evidence of viral pneumonia or hypoxia.
  Interventions: Other: Physical Activity Level; Other: Anxiety and Depression Assessment; Diagnostic Test: Exercise Capacity; Diagnostic Test: Pulmonary Function Test; Diagnostic Test: Cardiopulmonary Fitness Level; Other: Cognitive Assessment
- Pneumonia: Patients with clinical signs of pneumonia (fever, cough, dyspnoea, fast breathing) but no signs of severe pneumonia, including SpO2 ≥ 90% on room air
  Interventions: Other: Physical Activity Level; Other: Anxiety and Depression Assessment; Diagnostic Test: Exercise Capacity; Diagnostic Test: Pulmonary Function Test; Diagnostic Test: Cardiopulmonary Fitness Level; Other: Cognitive Assessment
- Severe Pneumonia: Patients with clinical signs of pneumonia (fever, cough, dyspnoea,fast breathing) plus one of the following: respiratory rate > 30 breaths/min; severe respiratory distress; or SpO2 < 90% on room air.
  Interventions: Other: Physical Activity Level; Other: Anxiety and Depression Assessment; Diagnostic Test: Exercise Capacity; Diagnostic Test: Pulmonary Function Test; Diagnostic Test: Cardiopulmonary Fitness Level; Other: Cognitive Assessment
- Critical Disease: Patients have one of the following: acute respiratory distress syndrome; sepsis; or septic shock.
  Interventions: Other: Physical Activity Level; Other: Anxiety and Depression Assessment; Diagnostic Test: Exercise Capacity; Diagnostic Test: Pulmonary Function Test; Diagnostic Test: Cardiopulmonary Fitness Level; Other: Cognitive Assessment

INTERVENTIONS:
Other: Physical Activity Level — International Physical Activity Questionnaire
Other: Anxiety and Depression Assessment — Hospital Anxiety and Depression Scale
Diagnostic Test: Exercise Capacity — 6 Minute Walk Test
Diagnostic Test: Pulmonary Function Test — Spirometry
Diagnostic Test: Cardiopulmonary Fitness Level — Cardiopulmonary Exercise Test
Other: Cognitive Assessment — Montreal Cognitive Assessment

SUMMARY:
COVID-19 (Coronavirus disease 2019) is a new infectious disease caused by a virus named as SARS-CoV2 (Severe Acute Respiratory Syndrome Coronavirus-2). Although it can have a devastating effect on many organs, the respiratory tract is particularly affected. In the course of the disease, a wide clinical spectrum is observed, from flu-like illness to lung failure. Some of the patients who survived the disease continue to have problems such as shortness of breath, fatigue, decrease in walking distance, decrease in participation in daily life activities. These problems suggest that the effects on respiratory and cardiac functions continue even after the disease ends. This study was designed to demonstrate the effects and extent of COVID-19 on cardiopulmonary capacity.

DETAILED DESCRIPTION:
Aims of the research are that demonstrate change in cardiopulmonary fitness level in patients with COVID-19 according to normal values and reveal the relationship of this change with age, gender, physical activity level, disease severity and accompanying medical conditions.

Patients older than 18 years old who are diagnosed with COVID-19 according to clinical symptoms and rt-PCR test positivity and at least 30 days past the end of their symptoms are accepted for the study.

According to World Health Organization's (WHO) classification, COVID-19 disease severity is determined. Physical activity level of the patients before COVID-19 is evaluated with International Physical Activity Questionnaire. Risk of anxiety and depression of the patients is identified with Hospital Anxiety and Depression Scale (HADS), which has 14 questions. To evaluate cardiopulmonary fitness level, cardiopulmonary exercise test (CPET) and 6-minute walk test are applied. Cardiopulmonary exercise test is gold standard to determine cardiac and respiratory functions. Pulmonary function test is performed to identify the conditions that affect the results of cardiopulmonary exercise test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SARS-Cov2 with a positive result of reverse polymerase-transcriptase chain reaction test
* It must have been at least 30 days after symptoms of COVID-19 improved.

Exclusion Criteria:

* 5 days after acute myocardial infarction
* Unstable angina
* Active endocarditis, myocarditis or pericarditis
* Symptomatic severe aortic stenosis
* Uncontrolled heart failure
* Acute pulmonary embolus, pulmonary infarction or thrombosis of lower extremities
* Suspected dissecting aneurysm
* Uncontrolled asthma
* Room air desaturation at rest (O2 ⩽85%)
* Respiratory failure
* Acute non-cardiopulmonary disorder that may affect exercise performance or be aggravated by exercise
* Mental impairment
* Severe untreated arterial hypertension at rest (>200 mm Hg systolic, >120 mm Hg diastolic)
* High-degree atrioventricular block
* Orthopaedic, neurological or systemic impairments that leading to inability to perform test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients applying to COVID-19 follow-up clinics
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen uptake | 1-6 months
  Cardiopulmonary exercise test
Oxygen uptake at anaerobic threshold | 1-6 months
  Cardiopulmonary exercise test
Borg rating of perceived exertion scale | 1-6 months
  Cardiopulmonary exercise test
Walk distance | 1-6 months
  6 minute walk test

SECONDARY OUTCOMES:
Borg dyspnea scale | 1-6 months
  Cardiopulmonary exercise test
Anxiety score | 1-6 months
  Hospital Anxiety and Depression Scale
Depression score | 1-6 months
  Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Faculty of Medicine, Physical Medicine and Rehabilitation Department, Ankara, Turkey (Türkiye)